CLINICAL TRIAL: NCT03689361
Title: Interest of the T2 * Sequence in MRI for the Diagnosis of Migraine Aura in the Acute Phase.
Acronym: MARIE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: RC31/16/8249; 2017-004091-60 (EudraCT Number)
Record Dates: First submitted 2018-09-20; First posted 2018-09-28 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: Migraine Aura
Keywords: migraine aura
MeSH Terms: conditions — Migraine with Aura

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- with migraine aura. (Other): patient with migraine aura detected by MRI, then MRI control 3 month after
  Interventions: Combination Product: MRI; Diagnostic Test: MRI control
- without migraine aura (Other): patient without migraine aura detected by MRI, then telephone consultation 3 month after
  Interventions: Other: telephone consultation

INTERVENTIONS:
Combination Product: MRI — Routine MRI with all the sequences performed for the management of acute neurological deficit in the Toulouse Neuro Vascular Unit (diffusion, FLAIR, T2 *, vascular sequences (AngioRM and TOF) and perfusion).
  Arms: with migraine aura.
Diagnostic Test: MRI control — MRI with all the sequences performed for the management of acute neurological deficit in the Toulouse Neuro Vascular Unit (diffusion, FLAIR, T2 *, vascular sequences (AngioRM and TOF) and perfusion)
  Arms: with migraine aura.
Other: telephone consultation — telephone consultation
  Arms: without migraine aura

SUMMARY:
investigators hypothesize that T2 * vein abnormalities are frequent and are specific to the migraine aura.

DETAILED DESCRIPTION:
The diagnosis of migraine aura is now based solely on clinical criteria and the assertion of the diagnosis on these clinical criteria alone proves difficult in the acute phase. Added to this difficulty, the symptomatology of a migraine aura can sometimes be similar to that of a stroke, so a diagnosis can be poorly established, resulting in poor patient care. The possibility of making the positive diagnosis of migraine aura on a routine MRI sequence, T2 *, would be an important advance for the management of these patients

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 55 years
* Admitted to the Neuro-Vascular Intensive Care Unit for Acute Focused Neurological Symptoms and MRI

  * less than 4 hours 30 minutes after onset of symptoms if symptoms persist during admission
  * less than two hours after the disappearance of symptoms if the patient arrives asymptomatic
* Affiliated to a social protection scheme.
* Having given their informed consent

Exclusion Criteria:

* Patients with neurological signs pointing to vertebrobasilar localization (vertigo, diplopia) or with a disorder of consciousness
* Presence of recent explanatory abnormalities on the MRI to make a diagnosis compatible with the initial neurological symptomatology (visible stroke in diffusion, cerebral hemorrhage, tumor, arteriovenous malformations).
* Potential strong cause of stroke known or discovered at the arrival of the patient, in particular stenosis of a cervical or intracranial artery upstream of the cerebral zone may correspond to the symptoms and emboligenic heart disease type atrial fibrillation.
* Pregnant women - Patients with a contraindication for MRI.
* Patients benefiting from a system of legal protection (tutelage,

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2018-12-22 (Actual); Primary Completion 2020-10-11 (Actual); Study Completion 2020-12-11 (Actual)

PRIMARY OUTCOMES:
frequency of the presence of visible brain vein abnormalities | Day 0
  visible brain vein abnormalities on T2 * sequences MRI ,

SECONDARY OUTCOMES:
perfusion parameters | Day 0
  in MRI , Overall visual assessment: presence or absence of hypoperfusion (presence or not in each anterior, middle and posterior territory) each lobe: Frontal, Temporal, Parietal, Occipital)
asymmetry of visualization of the 3 intracranial arteries in MRI | Day 0
  in MRI TOF

CONTACTS AND LOCATIONS:
Overall Officials: Alain Viguier, PH, Principal Investigator — Uuniversity Hospital Toulouse
Locations (1):
- Hôpital Pierre Paul Riquet - CHU de Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No